CLINICAL TRIAL: NCT03880773
Title: Tri Stapler vs. Ultrasonic Scalpel in Distal Pancreatectomy
Brief Title: Comparison Between Two Methods of Pancreatic Transection in Distal Pancreatectomy
Acronym: TRUDY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRUDY
Record Dates: First submitted 2019-02-25; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Fistula; Distal Pancreatectomy
MeSH Terms: conditions — Pancreatic Fistula | interventions — Surgical Staplers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stapler (Experimental)
  Interventions: Device: Stapler
- ultrasonic shears (Active Comparator)
  Interventions: Device: ultrasonic shears

INTERVENTIONS:
Device: Stapler — for transection of the pancreas and pancreatic stump treatment
  Arms: Stapler
Device: ultrasonic shears — for transection of the pancreas and pancreatic stump treatment
  Arms: ultrasonic shears

SUMMARY:
Several systematic reviews have investigated the management of the pancreatic stump in order to reduce the postoperative pancreatic fistula (POPF) rate after distal pancreatectomy (DP). The appropriate closure technique of the pancreatic stump is still debated. There is no published experience about the comparison of the Endo GIA Reinforced Reload with Tri-Staple Technology (TS) versus Harmonic Focus (US) after distal pancreatectomy (DP) regarding the reduction of POPF.

The investigators want to compare the incidence of clinically-relevant POPF (CR-POPF) after DP, depending upon the transection technique (TS versus US).

This is a randomized controlled, multicenter, patient-blinded, superiority trial. This protocol was designed according to the SPIRIT guidelines.

Two groups of 76 patients (152 in total) with an indication for elective minimally invasive or open DP for a lesion of the body-tail of the pancreas. The two techniques analyzed are Endo GIA Reinforced Reload with Tri-Staple Technology (TS) and Harmonic Focus (US) as control.

The primary endpoint is to evaluate the incidence of CR-POPF rate after DP. Secondary endpoints are intraoperative outcomes (blood loss, operative time and conversion of the minimally invasive procedure), postoperative outcomes (complications rate; hospitalization parameters to 90 days; mortality) and treatment costs.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective DP via a minimally invasive (laparoscopic or robotic) or open technique, either preserving the spleen or with splenectomy, depending on the diagnosis/nature of the tumor
* ASA score < 4
* Ability of the subject to understand character and individual consequences of the clinical trial
* Written informed consent

Exclusion Criteria:

* Pancreas thickness >17mm measured at the intraoperative ultrasound at the pancreatic transection level
* Metastatic disease
* Kidney or adrenal gland resection
* Arterial resection (celiac axis, superior mesenteric artery, hepatic artery)
* Intestinal resections and anastomoses or stoma
* Acute necrotizing and chronic pancreatitis
* Immune suppressed patients
* Pregnant women
* Patients with contraindications for distal pancreatectomy
* Impaired mental state or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Pancreatic fistula | 90 days
  pancreatic fistula according to International Study Group of Pancreatic Surgery (ISGPS) 2017 definition

SECONDARY OUTCOMES:
Operative time | intra-operatively
Rate of postoperative overall and specific complications | 30 days, 90 days
  abdominal collections, delayed gastric emptying, hemorrhage, sepsis, wound infections
Rate of re-operations or percutaneous drainage | 30 days, 90 days
  re-operations rate or percutaneous drainage rate
Cost-analysis | 90 days
  intra and post-operative costs

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Policlinico GB Rossi, Verona, Italy

REFERENCES:
- [Background] Ban D, Shimada K, Konishi M, Saiura A, Hashimoto M, Uesaka K. Stapler and nonstapler closure of the pancreatic remnant after distal pancreatectomy: multicenter retrospective analysis of 388 patients. World J Surg. 2012 Aug;36(8):1866-73. doi: 10.1007/s00268-012-1595-z. PMID 22526040
- [Background] Suzuki Y, Fujino Y, Tanioka Y, Hori Y, Ueda T, Takeyama Y, Tominaga M, Ku Y, Yamamoto YM, Kuroda Y. Randomized clinical trial of ultrasonic dissector or conventional division in distal pancreatectomy for non-fibrotic pancreas. Br J Surg. 1999 May;86(5):608-11. doi: 10.1046/j.1365-2168.1999.01120.x. PMID 10361178
- [Background] Kleeff J, Diener MK, Z'graggen K, Hinz U, Wagner M, Bachmann J, Zehetner J, Muller MW, Friess H, Buchler MW. Distal pancreatectomy: risk factors for surgical failure in 302 consecutive cases. Ann Surg. 2007 Apr;245(4):573-82. doi: 10.1097/01.sla.0000251438.43135.fb. PMID 17414606
- [Background] Knaebel HP, Diener MK, Wente MN, Buchler MW, Seiler CM. Systematic review and meta-analysis of technique for closure of the pancreatic remnant after distal pancreatectomy. Br J Surg. 2005 May;92(5):539-46. doi: 10.1002/bjs.5000. PMID 15852419
- [Background] Diener MK, Seiler CM, Rossion I, Kleeff J, Glanemann M, Butturini G, Tomazic A, Bruns CJ, Busch OR, Farkas S, Belyaev O, Neoptolemos JP, Halloran C, Keck T, Niedergethmann M, Gellert K, Witzigmann H, Kollmar O, Langer P, Steger U, Neudecker J, Berrevoet F, Ganzera S, Heiss MM, Luntz SP, Bruckner T, Kieser M, Buchler MW. Efficacy of stapler versus hand-sewn closure after distal pancreatectomy (DISPACT): a randomised, controlled multicentre trial. Lancet. 2011 Apr 30;377(9776):1514-22. doi: 10.1016/S0140-6736(11)60237-7. PMID 21529927
- [Background] Zhang H, Zhu F, Shen M, Tian R, Shi CJ, Wang X, Jiang JX, Hu J, Wang M, Qin RY. Systematic review and meta-analysis comparing three techniques for pancreatic remnant closure following distal pancreatectomy. Br J Surg. 2015 Jan;102(1):4-15. doi: 10.1002/bjs.9653. Epub 2014 Nov 12. PMID 25388952
- [Background] Kim H, Jang JY, Son D, Lee S, Han Y, Shin YC, Kim JR, Kwon W, Kim SW. Optimal stapler cartridge selection according to the thickness of the pancreas in distal pancreatectomy. Medicine (Baltimore). 2016 Aug;95(35):e4441. doi: 10.1097/MD.0000000000004441. PMID 27583852
- [Background] Peng YP, Zhu XL, Yin LD, Zhu Y, Wei JS, Wu JL, Miao Y. Risk factors of postoperative pancreatic fistula in patients after distal pancreatectomy: a systematic review and meta-analysis. Sci Rep. 2017 Mar 15;7(1):185. doi: 10.1038/s41598-017-00311-8. PMID 28298641